CLINICAL TRIAL: NCT01624753
Title: Clinical Utility of Fibered Confocal Fluorescence Microscopy Imaging in Patients With Diffuse Parenchymal Lung Diseases
Brief Title: Fibered Confocal Fluorescence Microscopy Imaging in Patients With Diffuse Parenchymal Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/245/Cfcfm
Record Dates: First submitted 2012-05-15; First posted 2012-06-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Parenchymal Lung Diseases
Keywords: interstitial lung disease; interstitial pneumonia; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- confocal microscopy (Experimental): During bronchoscopy, one side of the bronchial tree will be examined (either right or left) and targeted based on pre-procedure HRCT/CT scan findings. A 1.4mm diameter Alveoflex Confocal MiniprobeTM (MaunaKea Technologies, France) will be deployed down the working channel of the standard bronchoscope and advanced distally into the alveoli. Images are acquired by gentle contact providing real-time imaging and microstructural detail of the alveolus which will be continuously recorded during the procedure and stored for further morphometric and cellular analyses. Up to 10 bronchoalveolar areas will be observed and the location of the corresponding lung segment will be registered according to the international bronchial nomenclature.
  Interventions: Device: confocal microscopy

INTERVENTIONS:
Device: confocal microscopy — During bronchoscopy, one side of the bronchial tree will be examined (either right or left) and targeted based on pre-procedure HRCT/CT scan findings. A 1.4mm diameter Alveoflex Confocal MiniprobeTM (MaunaKea Technologies, France) will be deployed down the working channel of the standard bronchoscope and advanced distally into the alveoli. Images are acquired by gentle contact providing real-time imaging and microstructural detail of the alveolus which will be continuously recorded during the procedure and stored for further morphometric and cellular analyses. Up to 10 bronchoalveolar areas will be observed and the location of the corresponding lung segment will be registered according to the international bronchial nomenclature.
  Other Names: Fibered confocal fluorescence microscopy imaging; alveoloscopy; Alveoflex Confocal MiniprobeTM

SUMMARY:
Fibered confocal fluorescence microscopy (FCFM) (CellvizioR Lung, MaunaKea Technologies, France) could potentially provide diagnostic information on fibrosis and inflammation of the distal air spaces associated with diffuse parenchymal lung diseases without the need for lung biopsies, thereby fulfilling the gap in the investigators current medical practice of a minimally invasive procedures with few complications and a high diagnostic fidelity.

In patients scheduled for bronchoscopy as part of regular clinical care/diagnostic workup, the investigators will offer the patient concurrent FCFM imaging to be performed during the bronchoscopic procedure. The investigators aim to identify and catalogue distinct and discriminating features seen on images obtained from fibered confocal fluorescence microscopy in this group of patients, and to correlate these findings with specific high resolution computed tomography (HRCT) features and pathological findings if available. Eventually the investigators hope to create diagnostic criteria for fibered confocal fluorescence microscopy image interpretation of specific diffuse parenchymal lung disease entities.

DETAILED DESCRIPTION:
Diffuse parenchymal lung diseases (DPLD) represent a large and heterogeneous group of disorders encompassing a collection of pulmonary diseases that affect the interstitium including the alveolar epithelium, pulmonary capillary endothelium, basement membrane, perivascular and perilymphatic tissues. This spectrum of disease is encountered not only in pulmonary medicine as a collection of idiopathic conditions, but also in transplant medicine (solid organ and haematological), infectious disease (atypical pneumonias) and rheumatology (connective tissue disease/vasculitis). Although new techniques such as high resolution computed tomography (HRCT) and insights into the pathogenesis have led to a better understanding of DPLD, clinical diagnosis, management and prognostication remains a challenge.

The current diagnostic standard of DPLD is a correlation between clinical course, radiological features on HRCT and pathological findings. Even in idiopathic pulmonary fibrosis (IPF) where a typical usual interstitial pattern on HRCT is pathognomonic without the requirement of pathology, this is only diagnostic in 80% of patients, and an atypical pattern on HRCT does not preclude a diagnosis of IPF. As such the final diagnosis often hinges on histopathological confirmation which traditionally requires a surgical lung biopsy under general anaesthetic via thoracoscopy or thoracotomy. This entails significant morbidity and mortality in this group of patients who already have respiratory compromise. Minimally invasive endoscopic procedures such as bronchoalveolar lavage (BAL) and transbronchial lung biopsy (TBLB) via flexible bronchoscopy have increasingly been used in the majority of cases as a substitute to surgical biopsy. This unfortunately is not entirely a benign procedure either - BAL can worsen hypoxaemia, and TBLB may lead to significant bleeding or pneumothorax in around 5% of patients. Furthermore, the diagnostic yield of TBLB is severely limited because of the small size of tissue and the blind nature of choosing target bronchopulmonary segments to biopsy. Other limitations include significant inter-observer variation in interpretation of the histology, and the problem of ''sampling error'': the possibility that a biopsy specimen was taken from an area not representative of the predominant disease process. These limitations are reflected in the low diagnostic yields reported - in immunocompromised patients, the diagnostic yield of either BAL or TBLB was 38% with a 13% complication rate, and diagnostic yields of <50% with TBLB have been reported in hypersensitivity pneumonitis and about 30% in usual interstitial pneumonia.

A definitive diagnosis is essential in the management of diffuse parenchymal lung diseases. Infectious aetiologies necessitate antimicrobial therapy while immune mediated causes are managed by immunosuppression. Drug induced pathology will require a revision of current medication while fibrotic conditions can be managed expectantly. Prognostication is also markedly altered by aetiology and diagnosis. The gap in current medical practice is the availability of minimally invasive procedures with few complications and a high diagnostic fidelity.

Fibered confocal fluorescence microscopy (FCFM) (CellvizioR Lung, MaunaKea Technologies, France) is a new, safe and minimally invasive technique that can be used to obtain real time high-resolution, microstructural images of lobular and alveolar lung structures in living humans. FCFM provides a clear, in-focus image of a thin section within a biological sample, where the microscope's objective is replaced by a flexible fiberoptic miniprobe. The technique makes it possible to obtain high-quality images from endogenous or exogenous tissue fluorophores, through a fiberoptic probe of 1.4mm diameter that can be introduced into the working channel of a standard, flexible bronchoscope. This could potentially provide diagnostic information on fibrosis and inflammation of the distal air spaces associated with diffuse parenchymal lung diseases without the need for lung biopsies.

Current data and imaging for pulmonary FCFM is available in normal alveoli of both smokers and non-smokers. Pathological lung FCFM imaging for DPLD has yet to be published. In patients scheduled for bronchoscopy as part of regular clinical care/diagnostic workup, the investigators will offer the patient concurrent fibered confocal fluorescence microscopy imaging to be performed during the bronchoscopic procedure. The investigators aim to identify and catalogue distinct and discriminating features seen on images obtained from FCFM in this group of patients, and to correlate these findings with specific HRCT features and pathological findings if available. The investigators hope to be able to demonstrate reproducibility of FCFM image interpretation, with minimal intra and inter observer variability and high Kappa values. Eventually the investigators hope to define diagnostic criteria and patterns for FCFM image interpretation to correlate with specific DPLD entities, thereby creating an atlas of FCFM for DPLD. This would enhance our current diagnosis and management of DPLD with minimal additional risks to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21 years old and older diagnosed with suspected diffuse parenchymal lung disease (multi-lobar pulmonary infiltrates)
2. Patients scheduled for bronchoscopy as part of regular clinical care/diagnostic workup
3. Ability and willingness to sign informed consent

Exclusion Criteria:

1. Contraindications to bronchoscopic evaluation eg. Haemodynamic instability, respiratory failure, uncorrected coagulopathy
2. Suspected/confirmed pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Univariate and multivariate logistic regression analysis of the FCFM image features identified to discriminate against HRCT features and pathology. | 5 years

SECONDARY OUTCOMES:
Utilize receiver operating characteristic (ROC) curves to identify the FCFM image feature or combination of features which demonstrates the best sensitivity and specificity for each HRCT feature and pathology. | 5 years
Comparison of the areas under the curves for the interpretation of 2 still FCFM image frames of the same sequence recording of a single alveolar segment. | 5 years
Using Kappa values to quantify a high study agreement (kappa >0.8) between the assessors and within an assessor for FCFM image interpretation. | 5 years
Complication rate of fibered confocal fluorescence microscopy over and above standard bronchoscopy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Su Ying Low, BMBCh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Thiberville L, Salaun M, Lachkar S, Dominique S, Moreno-Swirc S, Vever-Bizet C, Bourg-Heckly G. Human in vivo fluorescence microimaging of the alveolar ducts and sacs during bronchoscopy. Eur Respir J. 2009 May;33(5):974-85. doi: 10.1183/09031936.00083708. Epub 2009 Feb 12. PMID 19213792
- [Background] Thiberville L, Moreno-Swirc S, Vercauteren T, Peltier E, Cave C, Bourg Heckly G. In vivo imaging of the bronchial wall microstructure using fibered confocal fluorescence microscopy. Am J Respir Crit Care Med. 2007 Jan 1;175(1):22-31. doi: 10.1164/rccm.200605-684OC. Epub 2006 Oct 5. PMID 17023733
- [Background] Newton RC, Kemp SV, Yang GZ, Elson DS, Darzi A, Shah PL. Imaging parenchymal lung diseases with confocal endomicroscopy. Respir Med. 2012 Jan;106(1):127-37. doi: 10.1016/j.rmed.2011.09.009. Epub 2011 Oct 14. PMID 22000588